## **Cover Page for Statistical Analysis Plan**

| Sponsor-Investigator: | Spyridon Fortis |
|-----------------------|----------------------------------|
| NCT Number: | NCT03959982 |
| Unique Protocol ID: | 201905817 |
| Official Title: | The Effect of Heated, Humidified |
| | High-flow Air in COPD Patients |
| | With Chronic Bronchitis |
| Date of Document: | 01 July 2019 |

Assessment of the effectiveness of the intervention by assessing the change in the PSQI, CAT, and the 6-minute walk from enrollment to the 6-week visit. The Wilcoxon rank-sum test will be used to compare changes in PSQI, CAT, and the 6-minute walk test from enrollment to the 6-week visit between the intervention and the control group. The Wilcoxon rank-sum test will be used because the dependent variables will most likely not follow normal distribution.